CLINICAL TRIAL: NCT06319430
Title: The Role of Technology in Facilitating Play for Children With Physical Disabilities: Development of the Dice Model of Play
Brief Title: Technology in Play for Children With Physical Disabilities: the Dice Model of Play
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Rehabilitation Centre for Children, Canada (Other)
Responsible Party: Principal Investigator, Minoo Dabiri Golchin, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HS26236(H2023:343)
Record Dates: First submitted 2024-02-21; First posted 2024-03-20 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Disability Physical; Disabilities Mental
Keywords: play and playthings; Assistive technology; Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: The primary purpose is validation of..........
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robots (Experimental): Participants will be randomly allocated to groups A or B. Those in group A will co-design and build their LEGO™ robot, using the researcher's assistance, as led by the child. A go-along interview will be conducted during the co-design with the child . The co-design session will be video recorded to provide context, visual data, and to inform the qualitative analysis. Videos will be deleted right after analysis. A research assistant (RA) will visit the participant's home twice a week for 30 to 45 minutes (after school or on the weekend) to play with the child and their built LEGO™ robots for four weeks (4 sessions total).
  Interventions: Other: robots
- conventional toys (Experimental): Group B will engage in the same process of 4 play intervention sessions over four weeks with the research assistant; however, they will receive conventional play tools. The RA will carry a prepared play pack for the play intervention session.
  Interventions: Other: conventional

INTERVENTIONS:
Other: robots — LEGO robots with adaptation according to child's age and developmental skills.
  Arms: robots
Other: conventional — A pack of conventional play tools consists of dolls, teddy bears, miniature wild animals, and small cars. All are available, and the child can choose to play with them.
  Arms: conventional toys

SUMMARY:
Play is an important activity for children. Almost all children play, but what is play? It is not easy to define play. In the past, people believed that children played to burn their energy. Now, it is known that play is important for children's growth. Some kids with disabilities cannot play. Many experts use play to teach children specific skills. People often forget that play is a child's right. It is important to help all children play. The first step is to define play and find what features are important in helping a child with a disability play.

There are some models of play. But they are not complete. They do not look at play as a whole. Some models are just about playfulness, and some are about playing with others. Having a model that defines play helps researchers and clinicians think about play and the different parts of it. Then, when a child cannot play, experts can fix the part that is not working. Investigators want to introduce a model of play in this project. Investigators want to edit and complete it in three steps. First, Investigators will ask parents and children with disabilities about things that help or do not help them play; then, investigators will give Lego robots to kids that they will build with help and play with them for a few weeks. And at the end, investigators will ask therapists and other experts about our model of play. This model will be edited during the study.

DETAILED DESCRIPTION:
The study is designed in three phases, employing a mixed-method approach that integrates qualitative and quantitative methods. Phase 1 involves exploring the alignment of the Dice Model of Play with the experiences of 10 children (aged 3-8, diagnosed with different abilities) and their guardians through semi-structured interviews and content analysis; Phase 2 examines the practical application of the model with a cross-over design. Up to 20 children with different abilities will build their Lego robots within a co-design and will play with that robot for four sessions. The other group will play with conventional toys for four sessions. They will switch after finishing those sessions. Sessions will be directed by a master of occupational therapy student supervised by Dr. Jacquie Ripat, a registered occupational therapist in Manitoba. Assessments will be Test of Playfulness (TOP), enjoyment (PPE_DC), and play skills (ChIPPA-2) three times at the start, switching point, and last session. A go-along interview will be conducted in the co-design. Lastly, Phase 3 seeks expert opinions on the revised Dice Model of Play's clarity, relevance, and applicability, using online focus groups with professionals in occupational therapy, psychology, and computer science. The study aims to modify and enhance the model based on the findings from these phases.

ELIGIBILITY:
Inclusion Criteria:

* Having a disability or typically developed
* Between 3 to 8 years old
* Speaking and understanding English or Persian
* Living in Winnipeg

Exclusion Criteria:

* Not receiving play therapy within the last three months

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Test of Playfulness | before the session 1, after session 8, after session 16, each time 10 to 20 minutes.
  The Test of playfulness (TOP) version 4 (Bundy, 1998) is an observational test that covers four main elements of playfulness: intrinsic motivation, internal control, freedom of reality, and framing within 29 Likert scale related to extent, intensity, and skillfulness and is used for children between 15 months and 18 years old. Upper scores means better play skills, no cut-off score.
The Child Initiated Pretend Play Assessment (ChIPPA-2) | before the session 1, after session 8, after session 16, each time 18 minutes for 3 years old children and 30 minutes for 4-8 years old children.
  The Child Initiated Pretend Play Assessment (ChIPPA-2) provides a play tool pack consisting of two different sets: conventional and symbolic play tools. Percentage of Elaborated Play Actions (PEPA), Number of Object Substitutions (NOS), and Number of Imitations (NIA) are reported for conventional, symbolic, and general pretend play. Higher PEPA and NOS and lower NIA scores show better play skills. There are Z-scores for each age range that child can be compared with typically developed children.
The Pretend Play Enjoyment-Developmental Checklist (PPE-DC) | before the session 1, after session 8, after session 16, each time almost 10 minutes for parents and 10 minutes for researcher.
  The Pretend Play Enjoyment-Developmental Checklist (PPE-DC) measures play enjoyment and covers some aspects of pretend play, such as sequences, storytelling, playing with dolls, object substitution, roleplay, and social interaction, from parents and experts prospectives within two different scoresheets, items are defined for different developmental ages and by choosing one item, the play developmental age in each subcategory can be estimated. Play enjoyment score is better when is higher.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Centre for Children, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT06319430/Prot_SAP_ICF_000.pdf